CLINICAL TRIAL: NCT02155374
Title: Glucose Control for Glucocorticoid Induced Hyperglycemia During Chemotherapy
Acronym: GluCon-Chemo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Slotervaart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: NL47135.048.13
Record Dates: First submitted 2014-05-05; First posted 2014-06-04 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Hyperglycemia Steroid-induced
Keywords: Glucocorticoid induced hyperglycemia, insulin, chemotherapy
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin, Isophane; Isophane Insulin, Human; Nutrition Assessment; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sliding scale insulin (Active Comparator): Sliding scale insulin Glucose 7.8-12 mmol/l --> 2 IU insulin, glucose 12.1-17 mmol/l --> 4 IU insulin, glucose ≥17.1 mmol/l --> 6 IU insulin. In case of insufficient control, insulin doses will be increased
  Interventions: Drug: Sliding scale insulin; Behavioral: Dietary advice; Drug: Glucose lowering medication; Drug: Chemotherapy
- Intermediate acting insulin (Experimental): Intermediate acting insulin, 0.01 IU / mg prednison / kg body weight with a maximum of 0.5 unit insulin per kg body weight. In case of age > 70 years or diminished renal function (GFR <30ml/min)
  Interventions: Drug: Intermediate acting insulin; Behavioral: Dietary advice; Drug: Glucose lowering medication; Drug: Chemotherapy

INTERVENTIONS:
Drug: Sliding scale insulin
  Other Names: Short acting insulin on a sliding scale base
  Arms: Sliding scale insulin
Drug: Intermediate acting insulin
  Other Names: NPH insulin, insulatard
  Arms: Intermediate acting insulin
Behavioral: Dietary advice — Dietary advice to avoid food products with high glycemic index / high glucose load
Drug: Glucose lowering medication — Regular glucose lowering medication as prescribed by the patient's own physician before study entry
Drug: Chemotherapy — Chemotherapy (containing glucocorticoids) as prescribed by the patient's own physician
  Other Names: Antineoplastic therapy

SUMMARY:
Objective: to determine which regimen results in best glycemic control and safety profile, expressed as glucose values within target range and occurrence of hypoglycemia. Secondary objective is to compare patient satisfaction, clinical outcomes and toxicity.

Study design: Randomized open label cross-over study Study population: Patients ≥ 18 years, who developed glucocorticoid induced hyperglycemia requiring initiation or adjustment of antihyperglycemic agents in a previous chemotherapy cycle. Patient should have ≥2 cycles of chemotherapy scheduled, with 3-10 consecutive days of ≥12,5mg prednisone-equivalent glucocorticoid and a wash-out period of 4-38 days between each cycle.

Intervention: subjects will be treated by insulin regimen A and B in random order during two consecutive cycles of chemotherapy. A) intermediate acting insulin 0.01 IU / mg prednisone-equivalent / kg body weight once daily subcutaneous B) Short-acting insulin according to sliding scale regimen, dose adjusted to current grade of hyperglycemia.

Main study parameters: Difference in fraction of blood glucose measurements (BGM) within target range and occurrence of hypoglycemia.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Both study treatments are just a slight variation in regular care for glucocorticoid induced hyperglycemia. Glycemic control is likely to improve due to treatments and increased counselling. All subjects will receive both treatment regimens.

The burden consists of 16-32 extra BGMs over 2 x 4-10 days, wearing the glucose sensor, 1 venipuncture (if HbA1c and creatinin are not determined in routine laboratory within 3 months before start), and 1 randomization visit to the outpatient clinic. Potential risk is the occurrence of hypoglycemia, as is present in any insulin therapy. The investigators account for this risk by giving subjects dietary advice and education how to prevent, recognize and treat hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* Glucocorticoid induced hyperglycemia in previous cycle of chemotherapy that required therapy initiation or adjustment
* Duration of glucocorticoid cycles 3-10 consecutive days and 4-38 glucocorticoid-free days between 2 cycles
* Prednisone-equivalent dose of ≥ 12,5mg
* At least 2 more cycles of chemotherapy to receive

Exclusion Criteria:

* History of hypo-unawareness
* Continuous tube or parental feeding
* Continuous (maintenance) systemic glucocorticoid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 24h till end of treatment (expected duration 4-8 days)
  Compare achievement of glycemic control in SSI therapy and intermediate acting insulin. Glycemic control is measured as the proportion of blood glucose measurements (BGM) within target range in each subject after 24h of treatment

SECONDARY OUTCOMES:
Patient satisfaction | At the end of each treatment cycle (expected duration 4-8 days)
  Compare patient satisfaction in each treatment regimen at a 6-point Likert scale, in the last cycle we evaluate patient's preference for glucose lowering treatment in next chemotherapy cycle (SSI or intermediate acting insulin)
Clinical outcomes | During each treatment (expected duration 4-8 days)
  Difference in clinical outcomes: incidence of oral candidiasis, pooled incidence of grade 3-4 chemotoxicity. Data on clinical outcomes will be collected by taking the patient history at the end of each treatment cycle.
Hypoglycemia | During each treatment (expected duration 4-8 days)
  Incidence of hypoglycemia in each treatment cycle defined as an interstitial glucose ≤ 3.9 mmol/l continuing until the interstitial glucose is >3.9 mmol/l

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Slotervaart Hospital, Amsterdam
  - Antoni van Leeuwenhoek hospital, Amsterdam
  - Isala Clinics, Zwolle